CLINICAL TRIAL: NCT04023721
Title: A Phase 2, Exploratory Study Evaluating the Safety and Antiviral Efficacy of Inarigivir Soproxil in Non-cirrhotic, Hepatitis B e Antigen-negative Subjects Infected With Chronic Hepatitis B Virus and Receiving or Stopping Treatment With a Nucleoside/Nucleotide Inhibitor
Brief Title: Evaluating the Safety and Efficacy of Inarigivir in Non-cirrhotic, Hepatitis B e Antigen-negative Subjects Infected With HBV Virus and Receiving or Stopping Treatment With a NUC Inhibitor
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety
Sponsor: F-star Therapeutics, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBP-9200-HBV-206
Record Dates: First submitted 2019-06-21; First posted 2019-07-17 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis B; HBV; Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Nucleosides; Nucleotides; Nucleobindins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 - Inarigivir Soproxil Alone (Experimental): Cohort 1, 400 mg Inarigivir daily for 24 weeks and after treatment discontinuation will be followed for a further 18 months.
  Interventions: Drug: Inarigivir soproxil
- Cohort 2 Arm A - Inarigivir Soproxil and NUC (Experimental): Cohort 2, Arm A, 400 Inarigivir daily in addition to their prestudy nucleoside/nucleotide (NUC) analogue inhibitors for 48 weeks. At Week 48 subjects will stop both inarigivir and the NUC and be followed for a further 48 weeks off treatment.
  Interventions: Drug: Inarigivir soproxil; Drug: Nucleoside/nucleotide (NUC) analogue inhibitors
- Cohort 2 Arm B - Inarigivir Soproxil and NUC (Experimental): Cohort 2, Arm B, 400 mg Inarigivir daily plus prestudy nucleoside/nucleotide (NUC) analogue inhibitors for at least 24 weeks and up to 48 weeks. After treatment discontinuation of both inarigivir and the NUC, subjects will be followed off treatment up to Week 96.
  Interventions: Drug: Inarigivir soproxil; Drug: Nucleoside/nucleotide (NUC) analogue inhibitors

INTERVENTIONS:
Drug: Inarigivir soproxil — Inarigivir soproxil 200 mg tablets
Drug: Nucleoside/nucleotide (NUC) analogue inhibitors — Continuation of prestudy NUC therapy
  Arms: Cohort 2 Arm A - Inarigivir Soproxil and NUC; Cohort 2 Arm B - Inarigivir Soproxil and NUC

SUMMARY:
An open-label, Phase 2, exploratory study to examine the safety and efficacy of inarigivir in non-cirrhotic, hepatitis B e antigen (HBeAg)-negative subjects with chronic HBV infection.

ELIGIBILITY:
Inclusion Criteria:

1. HBV-infected male and female subjects aged 18 to 70 years, inclusive
2. Ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI) within 6 months of enrollment (Cohort 1) or randomization (Cohort 2) date with no evidence of cirrhosis or hepatocellular carcinoma (HCC)
3. Must be willing and able to comply with all study requirements
4. Have HBV DNA <LLOQ at Screening
5. ALT normal or, if elevated, <2× ULN with a documented etiology for elevation such as non-alcoholic fatty liver disease (NAFLD) confirmed by either ultrasound or controlled attenuation parameter (CAP) score >280 on elastography
6. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of IP. If the urine pregnancy test is positive, a follow-up serum test is required for confirmation
7. Women of childbearing potential must agree to use a highly effective method of contraception throughout the study and for 3 months after discontinuing study treatment. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception throughout the study and for 3 months after discontinuing study treatment. Male subjects must not donate sperm throughout the study and for 3 months after discontinuing study treatment.

   * Women of childbearing potential are sexually mature women who have not undergone bilateral tubal ligation, bilateral oophorectomy, or hysterectomy; or who have not been postmenopausal (ie, who have not menstruated at all) for at least 1 year.
   * Highly effective methods of contraception are hormonal contraceptives (oral, injectable, patch, intrauterine devices), male partner sterilization, or total abstinence from heterosexual intercourse, when this is the preferred and usual lifestyle of the subject. Note: The double-barrier method (eg, synthetic condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel), periodic abstinence (such as calendar, symptothermal, post-ovulation), withdrawal (coitus interruptus), lactational amenorrhea method, and spermicide only are not acceptable as highly effective methods of contraception.
8. Must have the ability to understand and sign a written informed consent form (ICF); consent must be obtained prior to initiation of study procedures

In addition, subjects must meet the cohort-specific criteria listed below:

Cohort 1:

1. HBeAg-negative subjects on documented NUCs for ≥3 years with undetectable HBV DNA by polymerase chain reaction (PCR) documented at least annually over the last 2 years. NUCs can include tenofovir, entecavir, telbivudine, lamivudine, adefovir, and tenofovir-5TC.
2. HBsAg <1000 IU at Screening
3. Planning to discontinue NUC therapy

Cohort 2:

1. HBeAg-negative subjects on documented NUCs for ≥1 year with undetectable HBV DNA by PCR documented on at least 1 occasion in the last 6 months. NUCs can include tenofovir, entecavir, telbivudine, lamivudine, adefovir, and tenofovir-5TC.
2. Planning to continue NUC therapy

Exclusion Criteria:

1. Any prior liver biopsy evidence of metavir F3 or F4 disease
2. Any history of decompensation of liver disease including history of ascites, encephalopathy, or varices
3. Evidence of advanced fibrosis as defined by Fibroscan at the Screening Visit of

   ≥8 kPa. If Fibroscan is not available, subjects with both a Fibrotest ≥0.65 and aspartate transaminase (AST):platelet ratio index (APRI) ≥1.0 are excluded (subjects will not be excluded if only 1 of the Fibrotest or APRI results is higher than allowed)
4. Laboratory parameters not within defined thresholds:

   4.1 White blood cells <4000 cells/μL (<4.0×109/L) 4.2 Hemoglobin <11 g/dL (<110 g/L) for females, <13 g/dL (<130 g/L) for males 4.3 Platelets <130,000 per μL (<130×109/L) 4.4 Albumin <3.5 g/dL (<35 g/L) 4.5 International normalized ratio (INR) >1.5 4.6 Total bilirubin >1.2 mg/dL (>20.52 μmol/L) or alpha-fetoprotein (AFP) >50 ng/mL (>180.25 nmol/L). Subjects with an elevated indirect bilirubin and known Gilbert's disease can be included if direct bilirubin is within normal limits. Subjects with an AFP >50 ng/mL but <500 ng/mL can be included if CT scan or MRI performed within 3 months shows no evidence of HCC 4.7 Creatinine >1.2 mg/dL (>106.08 μmol/L) and creatinine clearance <50 mL/min (<0.83 L/s/m2)
5. Co-infection with hepatitis C virus (HCV), human immunodeficiency virus (HIV), or hepatitis D virus
6. Evidence or history of HCC
7. Malignancy within 5 years prior to Screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible
8. Significant cardiovascular, pulmonary, or neurological disease
9. Received solid organ or bone marrow transplant
10. Received within 3 months of Screening or expected to receive prolonged therapy with immunomodulators (eg, corticosteroids) or biologics (eg, monoclonal antibody, IFN)
11. Subjects currently taking medication(s) that are transported through organic anion transporting polypeptide 1 (OATP1) including, but not limited to, atazanavir, rifampin, cyclosporine, eltrombopag, gemfibrozil, lopinavir/ritonavir, and saquinavir
12. Use of another investigational agent within 3 months of Screening
13. Current alcohol or substance abuse judged by the Investigator to potentially interfere with compliance
14. Females who are pregnant or may wish to become pregnant during the study
15. If the Investigator believes the prospective subject will not be able to comply with the requirements of the protocol and complete the study
16. Any medical condition that, in the opinion of the Investigator, could interfere with evaluation of the study objectives or safety of the subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects reporting an adverse event, clinically significant adverse event, or laboratory abnormality | 28 to 52 weeks
  Proportion of subjects in Cohort 1 and 2 reporting an adverse event, clinically significant adverse event, or laboratory abnormality from start to end of treatment, and 30 days after stopping treatment
Change in quantitative HBsAg (Cohort 1) | Baseline to Week 24
  Reduction in quantitative hepatitis B surface antigen (HBsAg) by >0.3 log10 from Baseline to Week 24 of subjects in Cohort 1
Change in the percentage of subjects with loss of HBsAg (Cohort 1) | Baseline to Weeks 24 and Week 48
  Percentage of subjects in Cohort 1 with loss of hepatitis B surface antigen (HBsAg) from Baseline to Weeks 24 and 48
Percentage of subjects with ALT flares (Cohort 1) | 96 Weeks
  Percentage of subjects in Cohort 1 with alanine transaminase (ALT) flares, defined as ALT >200 IU or hepatitis B virus (HBV) DNA >20,000 IU
Percentage of subjects with suppression of HBV DNA <2000 IU/L (Cohort 1) | Weeks 24
  Percentage of subjects in Cohort 1 with suppression of hepatitis B virus (HBV) DNA <2000 IU/L at Weeks 24 and 48
Percentage of subjects with suppression of HBV DNA <2000 IU/L (Cohort 1) | Weeks 48
  Percentage of subjects in Cohort 1 with suppression of hepatitis B virus (HBV) DNA <2000 IU/L at Weeks 24 and 48
Percentage of subjects with ALT <40 IU/L (Cohort 1) | Weeks 24
  Percentage of subjects in Cohort 1 with alanine transaminase (ALT) <40 IU/L at Weeks 24, 48, 72, and 96
Percentage of subjects with ALT <40 IU/L (Cohort 1) | Weeks 48
  Percentage of subjects in Cohort 1 with alanine transaminase (ALT) <40 IU/L at Weeks 24, 48, 72, and 96
Percentage of subjects with ALT <40 IU/L (Cohort 1) | Weeks 72
  Percentage of subjects in Cohort 1 with alanine transaminase (ALT) <40 IU/L at Weeks 24, 48, 72, and 96
Percentage of subjects with ALT <40 IU/L (Cohort 1) | Weeks 96
  Percentage of subjects in Cohort 1 with alanine transaminase (ALT) <40 IU/L at Weeks 24, 48, 72, and 96
Percentage of subjects who lose HBsAg (Cohort 1) | Weeks 72
  Percentage of subjects in Cohort 1 who lose hepatitis B surface antigen (HBsAg) at Weeks 72 and 96
Percentage of subjects who lose HBsAg (Cohort 1) | Weeks 96
  Percentage of subjects in Cohort 1 who lose hepatitis B surface antigen (HBsAg) at Weeks 72 and 96
Percentage of subjects with suppression of HBV DNA <2000 IU/L (Cohort 2) | Weeks 72
  Percentage of subjects in Cohort 2 with suppression of hepatitis B virus (HBV) DNA <2000 IU/L at Weeks 72 and 96 (off inarigivir treatment)
Percentage of subjects with suppression of HBV DNA <2000 IU/L (Cohort 2) | Weeks 96
  Percentage of subjects in Cohort 2 with suppression of hepatitis B virus (HBV) DNA <2000 IU/L at Weeks 72 and 96 (off inarigivir treatment)
Percentage of subjects with ALT <40 IU/L (Cohort 2 ) | Weeks 72
  Percentage of subjects in Cohort 2 with alanine transaminase (ALT) <40 IU/L at Weeks 72 and 96 (off inarigivir treatment)
Percentage of subjects with ALT <40 IU/L (Cohort 2 ) | Weeks 96
  Percentage of subjects in Cohort 2 with alanine transaminase (ALT) <40 IU/L at Weeks 72 and 96 (off inarigivir treatment)
Percentage of subjects with HBsAg <1000 IU (Cohort 2) | Weeks 72
  Percentage of subjects in Cohort 2 with alanine transaminase (ALT) <40 IU/L at Weeks 72 and 96 (off inarigivir treatment)
Percentage of subjects with HBsAg <1000 IU (Cohort 2) | Weeks 96
  Percentage of subjects in Cohort 2 with alanine transaminase (ALT) <40 IU/L at Weeks 72 and 96 (off inarigivir treatment)

SECONDARY OUTCOMES:
Change in serum levels of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 | Baseline to Week 96 (100 weeks)
  Fold change from Baseline in markers of innate immunity in serum of IFN-α, IFN-γ, TNF, IL-6, IL-10, and IP-10 in subjects in Cohort 1 and 2
Percentage of subjects with HBsAg decline >0.3 log10 (Cohort 2) | Weeks 12, 24, 48, 72, and 96
  Percentage of subjects in Cohort 2 with hepatitis B surface antigen (HBsAg) decline >0.3 log10 at Weeks 12, 24, 48, 72, and 96
Percentage of subjects with HBsAg decline >0.5 log10 (Cohort 2) | Weeks 12, 24, 48, 72, and 96
  Percentage of subjects in Cohort 2 with hepatitis B surface antigen (HBsAg) decline >0.5 log10 at Weeks 12, 24, 48, 72, and 96
Percentage of subjects with HBsAg loss (Cohort 2) | Weeks 24, 48, 72, and 96
  Percentage of subjects in Cohort 2 with hepatitis B surface antigen (HBsAg) loss at Weeks 24, 48, 72, and 96
Percentage of subjects with undetectable HBV DNA (Cohort 2) | Weeks 24, 48, 72, and 96
  Percentage of subjects in Cohort 2 with undetectable hepatitis B virus (HBV) DNA at Weeks 24, 48, 72, and 96
Percentage of subjects who suppress HBsAg <100 IU (Cohort 2) | Weeks 24, 48, 72, and 96
  Percentage of subjects in Cohort 2 who suppress hepatitis B surface antigen (HBsAg) <100 IU at Weeks 24, 48, 72, and 96
Change in serum HBV DNA, HBsAg, and HBV RNA in log10 IU/mL (Cohort 2) | Baseline to Week 96 (100 weeks)
  Change in serum hepatitis B virus (HBV) DNA, hepatitis B surface antigen (HBsAg), and HBV RNA in log10 IU/mL from Baseline to Weeks 12, 24, 48, 72, and 96 for subjects in Cohort 2

CONTACTS AND LOCATIONS:
Overall Officials: Don Mitchell, Study Director — Spring Bank Pharmaceuticals
Locations (7):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - GI Research Institute, Vancouver, British Columbia
  - LAIR Centre, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Liver Center, Toronto, Ontario
- United Kingdom (2):
  - Barts Health NHS Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England